CLINICAL TRIAL: NCT00000494
Title: Management of Patent Ductus in Premature Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 13; R01HL023121 (Other Grant/Funding Number: US NIH Grant Number)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2012-04

CONDITIONS: Cardiovascular Diseases; Defect, Congenital Heart; Ductus Arteriosus, Patent; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Defects, Congenital; Ductus Arteriosus, Patent; Heart Diseases | interventions — Indomethacin; Cardiovascular Surgical Procedures

INTERVENTIONS:
Drug: indomethacin
Procedure: surgery, cardiovascular

SUMMARY:
To evaluate the effects (up to one year of age) of indomethacin on the clinical course of patent ductus arteriosus (PDA) in premature infants (24 hours old or less) and to assess the relative merits of indomethacin and surgery in infants with persistent respiratory distress who were not treated early with indomethacin. Two concurrent trials were performed.

DETAILED DESCRIPTION:
BACKGROUND:

The incidence of patent ductus arteriosus is higher in premature infants than in full-term infants and is highest in premature infants who have respiratory distress syndrome. It is generally agreed that intervention in an asymptomatic infant with a small left-to-right shunt is unnecessary, since the patent ductus almost invariably closes spontaneously and thus does not require surgery. A few infants will demonstrate signs of a large shunt during the course of respiratory distress syndrome. Many of these infants will improve with medical management of congestive heart failure, but others require surgical closure. A third group of babies with respiratory distress have severe progressive pulmonary disease requiring ventilatory support. There was disagreement as to whether elimination of the patent ductus in these infants resulted in decreased mortality. A variety of therapeutic approaches was being used, and there was no convincing evidence of the superiority of one treatment over another.

DESIGN NARRATIVE:

Trial A was a randomized, double-blind trial in which indomethacin plus usual medical therapy was compared with a placebo plus medical therapy. Where this regimen was unsuccessful, the code was broken, and infants who received indomethacin were treated surgically. Infants who had received placebo in Trial A were entered, if there were no contraindications to indomethacin, into Trial B. In Trial B, infants were randomized to surgery or indomethacin therapy. Those in whom indomethacin treatment was unsuccessful were treated surgically. The Recruitment and Intervention Phase began in April 1979. All patients were enrolled by March 31, 1981, and followed for one year after enrollment.

ELIGIBILITY:
Boy and girl premature infants with patent ductus arteriosus. Birth weight of 1,750 grams or less. Admitted to participating institution within first 24 hours of life.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1978-09; Study Completion 1982-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Nadas — Children's Hospital & Medical Center

REFERENCES:
- [Background] Gersony WM, Peckham GJ, Ellison RC, Miettinen OS, Nadas AS. Effects of indomethacin in premature infants with patent ductus arteriosus: results of a national collaborative study. J Pediatr. 1983 Jun;102(6):895-906. doi: 10.1016/s0022-3476(83)80022-5. PMID 6343572
- [Background] Ellison RC, Peckham GJ, Lang P, Talner NS, Lerer TJ, Lin L, Dooley KJ, Nadas AS. Evaluation of the preterm infant for patent ductus arteriosus. Pediatrics. 1983 Mar;71(3):364-72. PMID 6338474
- [Derived] Irawati Y, Natalia MER, Gondhowiardjo TD, Dachlan I, Soebono H. Modified tarsorrhaphy versus gold weight implant technique for paralytic lagophthalmos treatment in patients with leprosy: One-year observation of a randomized controlled trial study. Front Med (Lausanne). 2023 Jan 4;9:941082. doi: 10.3389/fmed.2022.941082. eCollection 2022. PMID 36687442